CLINICAL TRIAL: NCT03214783
Title: A Case-control Study to Assess the Association Between Facial Characteristics and Coronary Artery Diseases
Status: Completed | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2017-907
Record Dates: First submitted 2017-07-08; First posted 2017-07-12 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Coronary Artery Disease
Keywords: artificial intelligence; facial recognition; facial characteristic
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Coronary artery disease (CAD) group: Patients enrolled with at least one coronary lesion stenosis ≥50% according to coronary computer tomography or coronary angiography will be assigned to CAD group.
  Interventions: Other: Facial characteristics
- No CAD group: Patients enrolled without coronary lesion stenosis ≥50% according to coronary computer tomography or coronary angiography will be assigned to CAD group.
  Interventions: Other: Facial characteristics

INTERVENTIONS:
Other: Facial characteristics — The exposures are facial characteristics which differ significantly in exposure rates between coronary artery disease (CAD) group and no CAD group.

SUMMARY:
The purpose of this study is to explore the facial characteristics associated with the increased risk of coronary artery diseases. The secondary purpose is to evaluate the diagnostic efficacy of appearance factors for coronary artery diseases.

DETAILED DESCRIPTION:
Several age-related appearance factors were described associated with increased risk of coronary artery diseases (CAD). However, several limitations made these facial risk factors hard to be utilized in clinical practice, including 1) low prevalence in CAD patients, 2) lack of specific definition, 3) poor reproducibility in artificial recognition.

Thus, we designed a case-control study to explore new, common and well-defined facial characteristics associated with CAD and evaluate the diagnostic efficacy of appearence factors in CAD. We will recuit 1150 patients with at least one coronary lesion stenosis ≥50% according to coronary angiography or coronary computer tomography (CAD group) and 1150 patients without coronary lesion stenosis≥ 50% (No CAD group) judged by coronary angiography or coronary computer tomography. We will collect patients' baseline information and facial images. One hand, we will explore the facial factors associated with CAD by comparing the exposure rates of different facial factors in CAD group and No CAD group based on artificial intelligence technology. On the other hand, we will build a CAD risk model based on facial factors, and evaluate the diagnostic effect of the model.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing coronary computer tomography or coronary angiography
* Written informed consent

Exclusion Criteria:

* Prior percutaneous coronary intervention (PCI)
* Prior coronary artery bypass graft (CABG)
* Without blood biochemistry outcome
* With artificially facial alteration (i.e. cosmetic surgery, facial trauma or make-up)
* Other situations which make patients fail to be photographed

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients who undergo coronary computer tomography or coronary angiography from both resident patients and outpatient.
Sampling Method: Non-Probability Sample
Enrollment: 2300 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
The association between facial factors and increased risk of coronary artery diseases | at the end of enrollment (6 months)

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital Chinese Academay of Medical Science and National Center for Cardiovascular Diseases, Beijing, Beijing Municipality, China